CLINICAL TRIAL: NCT02697955
Title: The Effect of Subsartorial Saphenous Block on Postoperative Pain Following Major Ankle and Hind Foot Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProtokolSB2
Record Dates: First submitted 2016-02-22; First posted 2016-03-03 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2016-09

CONDITIONS: Arthrosis; Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis | interventions — Drug Combinations; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine-epinephrine (Experimental): 10 mL of 5 mg/mL bupivacaine with 5 μg/mL epinephrine = 50 mg bupivacaine and 50 μg epinephrine
  Interventions: Drug: Bupivacaine-epinephrine
- Placebo (Placebo Comparator): 10 ml normal saline water (sodium chloride solution, 0,9%)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bupivacaine-epinephrine — 50 mg bupivacaine and 50 μg adrenalin
  Other Names: Marcain-adrenalin (combination drug); Marketing Authorisation Holder: AstraZeneca; Marketing Authorisation number: 10213
  Arms: Bupivacaine-epinephrine
Other: Placebo — 9 mg sodium chloride pr. ml (0,9 %)
  Other Names: Sodium chloride solution
  Arms: Placebo

SUMMARY:
The study investigates the effect of a ultrasound-guided subsartorial saphenous block on postoperative pain following major ankle and hind foot surgery.

DETAILED DESCRIPTION:
Major ankle and hind foot surgery causes intense postoperative pain. Implementation of continuous sciatic catheters has been a great success in reducing postoperative pain following these operations, but despite an effective sciatic catheter patients still report moderate to severe pain from the anteromedial side of the ankle. According to cadaver dissection studies the saphenous nerve innervates the anterior and medial parts of the ankle and talonavicular joint, and even though a saphenous block is standard procedure in many departments of anesthesiology worldwide, scientific evidence regarding the effect of the saphenous block on postoperative pain is lacking.

This study investigates the effect of a selective, ultrasound-guided subsartorial saphenous block on postoperative pain following major ankle and hind foot surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective ankle or hind foot surgery either: (1) total ankle arthroplasty, (2) ankle arthrodesis (3) subtalar arthrodesis or (4) triple arthrodesis
* Age ≥ 18
* American Society of Anaesthesiology Classification I-III
* Informed consent both orally and in writing after the patient has fully understood the protocol and its limitations.

Exclusion Criteria:

* Communication problems or dementia
* Allergies to any medical product used in the study
* Neuropathy of the sciatic or femoral nerve prior to the operation
* Morbus Charcot-Marie-Tooth disease, diabetic neuropathy, peripheral vascular disease
* Daily use of opioids
* Coagulation disorders
* Infection at the site of injection or systemic infection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Frequency of patients who experience significant pain at rest (change from no significant pain to significant pain) | Arrival at the Perioperative Section (within 30 minutes after surgery) and at t = 30 min, t = 45 min, t = 60 min, t = 75 min, t = 90 min, t = 105 min, t = 120. The beginning of the observation period (t0) is the registered time for the end of surgery.
  Pain scores evaluated using NRS (numeric rating scale). Significant pain is defined as NRS > 3 from the anterior and/medial side of the ankle joint. In case of significant pain, patients receive a rescue saphenous block with 10 ml bupivacaine-adrenaline.

SECONDARY OUTCOMES:
Sensory testing, infrapatellar branch (nociception is tested using a standardized Neuropen) | At the time point when the patients report a change to significant pain during the observation period. In case of no significant pain during the observation period, sensory testing is conducted at t = 120 min.
  Test of nociceptive response in the cutaneous innervation area of the infrapatellar branch (branch of the saphenous nerve). The test is performed in an area from the medial femoral condyle to the midline between the apex of patella and tibial tuberosity.
Sensory testing, sciatic nerve (nociception is tested using a standardized Neuropen) | Sensory test is conducted at arrival at the Perioperative Section (within 30 minutes after surgery)
  Test of nociceptive response in the sciatic cutaneous innervation area to confirm full sensory block of the sciatic nerve.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Fichtner Bendtsen, MD, phD, Study Director — Department of Anesthesiology, Aarhus University Hospital
Locations (1):
- Department of Anesthesiology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clendenen SR, Whalen JL. Saphenous nerve innervation of the medial ankle. Local Reg Anesth. 2013 Mar 6;6:13-6. doi: 10.2147/LRA.S42603. Print 2013. PMID 23630434
- [Background] Blumenthal S, Borgeat A, Neudorfer C, Bertolini R, Espinosa N, Aguirre J. Additional femoral catheter in combination with popliteal catheter for analgesia after major ankle surgery. Br J Anaesth. 2011 Mar;106(3):387-93. doi: 10.1093/bja/aeq365. Epub 2010 Dec 17. PMID 21169609
- [Background] White PF, Issioui T, Skrivanek GD, Early JS, Wakefield C. The use of a continuous popliteal sciatic nerve block after surgery involving the foot and ankle: does it improve the quality of recovery? Anesth Analg. 2003 Nov;97(5):1303-1309. doi: 10.1213/01.ANE.0000082242.84015.D4. PMID 14570643
- [Background] Chen J, Lesser J, Hadzic A, Resta-Flarer F. The importance of the proximal saphenous nerve block for foot and ankle surgery. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):372. doi: 10.1097/AAP.0b013e318295596a. No abstract available. PMID 23788076
- [Background] Kalthur SG, Sumalatha S, Nair N, Pandey AK, Sequeria S, Shobha L. Anatomic study of infrapatellar branch of saphenous nerve in male cadavers. Ir J Med Sci. 2015 Mar;184(1):201-6. doi: 10.1007/s11845-014-1087-2. Epub 2014 Feb 18. PMID 24535194
- [Background] Kerver AL, Leliveld MS, den Hartog D, Verhofstad MH, Kleinrensink GJ. The surgical anatomy of the infrapatellar branch of the saphenous nerve in relation to incisions for anteromedial knee surgery. J Bone Joint Surg Am. 2013 Dec 4;95(23):2119-25. doi: 10.2106/JBJS.L.01297. PMID 24306699
- [Background] Fisker AK, Iversen BN, Christensen S, Linde F, Nielsen KK, Borglum J, Bendtsen TF. Combined saphenous and sciatic catheters for analgesia after major ankle surgery: a double-blinded randomized controlled trial. Can J Anaesth. 2015 Aug;62(8):875-82. doi: 10.1007/s12630-015-0379-y. Epub 2015 Apr 8. PMID 25851020
- [Background] Bendtsen TF, Moriggl B, Chan V, Borglum J. Basic Topography of the Saphenous Nerve in the Femoral Triangle and the Adductor Canal. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):391-2. doi: 10.1097/AAP.0000000000000261. No abstract available. PMID 26079358
- [Derived] Bjorn S, Wong WY, Baas J, Nielsen KK, Borglum J, Hauritz RW, Bendtsen TF. The Importance of the Saphenous Nerve Block for Analgesia Following Major Ankle Surgery: A Randomized, Controlled, Double-Blind Study. Reg Anesth Pain Med. 2018 Jul;43(5):474-479. doi: 10.1097/AAP.0000000000000764. PMID 29667940